CLINICAL TRIAL: NCT05600790
Title: Mechanism of Mindfulness Based Online Intervention in Reducing Emotional Distress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xinghua Liu, Director, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20221107
Record Dates: First submitted 2022-10-24; First posted 2022-11-01 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Emotional Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the MIED+TAU group (Experimental): Intervention description: provide standard audio instructions for mindfulness exercises, introduce the nature and law of anxiety, depression and other emotions, the source of anxiety, depression and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Interventions: Behavioral: Mindfulness Intervention for Emotional Distress
- the TAU-only group (No Intervention): TAU consisted of all medicinal and psychological treatments received between baseline and follow-up (about five months). Medicinal treatments included receiving Lorazepam, Olanzapine, Paroxetine Hydrochloride, Sertraline, etc. Psychological treatments included receiving cognitive behavior therapy or psychodynamic therap

INTERVENTIONS:
Behavioral: Mindfulness Intervention for Emotional Distress — Mindfulness Intervention for Emotional Distress (MIED) program provide standard audio instructions for mindfulness exercises, introduce the nature and law of anxiety, depression and other emotions, the source of anxiety, depression and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Arms: the MIED+TAU group

SUMMARY:
This study hopes to:

1. explore whether, at the individual level, the improvement of mindfulness ability can promote peace of mind, reduce the frequency of mental wandering, weaken or cut off the cycle between negative mood and mind wandering, and improve the individual's attention monitoring ability and ability to engage in the present.
2. explore the impact of mindfulness intervention on intimate relationships in the eastern culture under the intimate relationship interaction model.
3. explore and propose the level of personality functioning could be a moderator of outcomes of MIED.

DETAILED DESCRIPTION:
Mind Wandering is the conscious experience when an individual's attention shifts from an ongoing task or external environment to an internal thought stream unrelated to tasks and external stimuli. Mind wandering is closely related to attention and emotion. Frequent mental wandering and negative emotions, especially depression and anxiety, are positively correlated (Smallwood et al., 2009). Mindfulness and mind wandering are essentially a state of consciousness. Trait mind wandering is a general tendency of individuals, representing the overall level of individual mind wandering. Mindfulness training can improve the level of mindfulness, and individuals are more involved in the present; This study hopes to explore whether, at the individual level, the improvement of mindfulness ability can promote peace of mind, reduce the frequency of mental wandering, weaken or cut off the cycle between negative mood and mind wandering, and improve the individual's attention monitoring ability and ability to engage in the present.

Some findings suggest that higher levels of mindfulness are associated with relationship outcomes between partners (Barnes, Brown, Krusemark, Campbell & Rogge, 2007). This paper aims to explore the impact of mindfulness intervention on intimate relationships in the eastern culture under the intimate relationship interaction model. The selected research objects were: emotionally troubled individuals who were not satisfied with the intimate relationship or marriage relationship, usually one of the parties in the intimate relationship, no matter male or female, no matter sexual orientation; The group received a 49-day Mindfulness Intervention for Emotional Distress (MIED), and the effect of detection.

Increasing evidence has demonstrated the positive effects of mindfulness-based interventions on a range of outcomes, including reducing depression and anxiety on a group level. However, rare research has identified who would most likely benefit from such interventions, especially when online mindfulness-based interventions have been popular, such as MIED in China. No consistent moderator has been found in terms of personal characteristics, including personal traits (de Vibe et al., 2015; Giluk, 2009; Hanley, 2016; Nyklíček & Irrmischer, 2017). While the level of personality functioning has been proposed by DSM-5 AMPD and ICD-11 as a dimensional criterion crossing normal personality and personality disorders (Bender, Morey & Skodol, 2011; Tyrer, Mulder, Kim, & Crawford, 2019), the current study proposes that it could be a moderator of outcomes of MIED. The results could help to explore the potential mechanism underlying the beneficial effects of the MIED theoretically and guide adaptations of MIED practically.

Experiential avoidance refers to individuals resisting experiences or trying to eliminate certain experiences (such as emotions, thoughts, physical feelings, memory and behavioral tendencies, etc.), and trying to adopt corresponding strategies to change these experiences and the situations in which the experiences are generated (Hayes, Wilson, Gifford, Follette, & Strosahl, 1996). Experiential avoidance has been proved to be a maintenance factor for many psychological disorders (Boelen & Reijntjes, 2008), and trying to hide or suppress unpleasant thoughts, feelings and physical feelings will increase the frequency and pain of these same experiences (Gross,1998; Gross,2002; Sloan, 2004; Wegner, 1994). According to some reviews, experiential avoidance is one of the beneficial effects of mindfulness (Brown, Bravo, Roos, & Pearson, 2015; Shapiro et al., 2006). However, at present, the measurement of experiential avoidance is limited to self-reported questionnaires, lacking objective measurement tools. Therefore, this study uses the dichotic listening task to measure experiential avoidance and explore the role of experiential avoidance as the effective mechanism of mindfulness intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with scores greater than 21 on the Kessler Psychological Distress Scale.

Exclusion Criteria:

* Subjects who could not access the Internet;
* Subjects with insufficient Chinese ability;
* Subjects who have participated in mindfulness based projects for more than 6 weeks before, and / or the current frequency of meditation practice is more than once a week;
* Patients with schizophrenia or psychotic affective disorder, current organic mental disorder, substance abuse disorder and generalized developmental disorder;
* Subjects at risk of suicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-10-29 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Weekly changes of Five Facet Mindfulness Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Five Facet Mindfulness Questionnaire is a self-reported questionnaire measuring mindfulness levels. Scores range from 39 to 195, with higher scores indicating higher levels of mindfulness.
Weekly changes of Patient Health Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Patient Health Questionnaire is a self-reported questionnaire measuring the degree of being troubled by various common physical symptoms. Scores range from 0 to 30.
  0~4 scores: no physical symptoms; 5~9 scores: mild physical symptoms; 10~14 scores: moderate physical symptoms; 15~30 scores: severe physical symptoms.
Weekly changes of Chinese Perceived Stress Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Chinese Perceived Stress Scale is a self-reported questionnaire measuring stress. Scores range from 0 to 56, with higher scores indicating higher levels of stress.
Weekly changes of 10-item Kessler Psychological Distress Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The 10-item Kessler Psychological Distress Scale is a self-reported questionnaire measuring distress. Scores range from 10 to 50, with higher scores indicating higher levels of distress.
Weekly changes of Overall Anxiety Severity and Impairment Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Overall Anxiety Severity and Impairment Scale is a self-reported questionnaire measuring anxiety. Scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
Weekly changes of Overall Depression Severity and Impairment Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Overall Depression Severity and Impairment Scale is a self-reported questionnaire measuring depression. Scores range from 0 to 20, with higher scores indicating higher levels of depression.
Weekly changes of Inner Peace Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Inner Peace Scale is a self-reported questionnaire measuring peace. Scores range from 0 to 28, with higher scores indicating higher levels of peace.
Weekly changes of Athens Insomnia Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Athens Insomnia Scale is a self-reported questionnaire measuring sleepy quality. Scores range from 0 to 24, with lower scores indicating higher levels of sleep quality.

SECONDARY OUTCOMES:
Moderation effect and possible changes of the Levels of Personality Functioning-Brief Form 2.0 during the intervention | pre-intervention; after the 3rd week intervention; after the 5rd week intervention; after the 7-week intervention
  The Levels of Personality Functioning-Brief Form 2.0 is a self-reported questionnaire measuring personality functioning. Scores range from 12 to 48, with higher scores indicating worse levels of personality functioning.
Moderation effect and possible changes of Personality Functioning Subscale of the Chinese Personality Organization Inventory during the intervention | pre-intervention; after the 3rd week intervention; after the 5rd week intervention; after the 7-week intervention
  Personality Functioning Subscale of the Chinese Personality Organization Inventory is a self-reported questionnaire measuring personality functioning. Scores range from 0 to 20, with higher scores indicating worse levels of personality functioning.
Weekly changes of Acceptance and Action Questionnaire-II during the first three weeks of intervention during the intervention | pre-intervention; after the 1st week intervention; after the 2nd week intervention; after the 3rd week intervention
  The Acceptance and Action Questionnaire-II is a self-reported questionnaire measuring experiential avoidance. Scores range from 7 to 49, with higher scores indicating higher levels of experiential avoidance.
Weekly changes of Interpersonal Mindfulness Scale during the intervention | pre-intervention; after the 3rd week intervention; after the 5rd week intervention; after the 7-week intervention
  The Interpersonal Mindfulness Questionnaire is a self-reported questionnaire measuring mindfulness level within interpersonal events, such as communication and emotion exchange. The 27-item scale contains four dimensions: focus on the present, awareness of self and others, non-judgmental acceptance, and non-reaction. Scores range from 0 to 135, with higher scores indicating higher levels of interpersonal mindfulness.
Weekly changes of Philadelphia Mindfulness Scale-Chinese Version during the intervention | pre-intervention; after the 3rd week intervention; after the 5rd week intervention; after the 7-week intervention
  Philadelphia Mindfulness Scale-Chinese Version is a self-reported questionnaire measuring awareness and acceptance levels. Scores range from 16 to 80, with higher scores indicating higher levels of awareness and acceptance.
Weekly changes of Attention-Related Cognitive Errors Scale during the intervention | pre-intervention; after the 3rd week intervention; after the 5rd week intervention; after the 7-week intervention
  Attention-Related Cognitive Errors Scale is a questionnaire for individuals to report the frequency of attention related cognitive errors. Scores range from 11 to 55, with higher scores indicating higher levels of the more mistakes occur without awareness.
Weekly changes of Mind-Wandering Questionnaire during the intervention | pre-intervention; after the 3rd week intervention; after the 5rd week intervention; after the 7-week intervention
  The Frequency of Mind Wandering Questionnaire is a self-reported scale for individual to evaluate the frequency of wandering. Scores range from 21 to 105, with higher scores indicating higher levels of mind wandering.
Weekly changes of Parter Acceptance Scale during the intervention | pre-intervention; after the 3rd week intervention; after the 5rd week intervention; after the 7-week intervention
  The Partner Acceptance Scale (PAS) is a self-reported questionnaire measuring one's acceptance level towards the other partner. Scores range from 0 to 35, with higher scores indicating higher levels of acceptancy.
Weekly changes of Test of Self-Conscious Affect-3 during the intervention | pre-intervention; after the 3rd week intervention; after the 5rd week intervention; after the 7-week intervention
  Test of Self-Conscious Affect-3 is a self-reported questionnaire measuring behavioral tendency of shame, guilt and etc. Scores range from 64 to 320, with higher scores indicating higher tendency of feeling certain self-conscious emotion.
Weekly changes of Brief Experiential Avoidance Questionnaire during the first three weeks of intervention | pre-intervention; after the 1st week intervention; after the 2nd week intervention; after the 3rd week intervention
  The Brief Experiential Avoidance Questionnaire is a self-reported questionnaire measuring experiential avoidance. Scores range from 15 to 90, with higher scores indicating higher levels of experiential avoidance.
Weekly changes of Couples Satisfaction Index during the intervention | pre-intervention; after the 3rd week intervention; after the 5rd week intervention; after the 7-week intervention
  The Couples Satisfaction Index (CSI) is a self-reported questionnaire measuring individual's subjective satisfaction towards couple. Scores range from 0 to 36, with higher scores indicating higher levels of satisfaction.
Weekly changes of the dichotic listening task during the first three weeks of intervention | pre-intervention; after the 1st week intervention; after the 2nd week intervention; after the 3rd week intervention
  The dichotic listening task is a computer-based behavioral task to measure experiential avoidance. The task involved presenting words into an unattending ear while worry or neutral scenarios were presented into the attending ear. Participants were given a surprise word recognition test of the words. Greater percentage of words recognition indicates higher levels of experiential avoidance.
Weekly changes of sustained attention response task during the intervention | pre-intervention; after the 3rd week intervention; after the 5rd week intervention; after the 7-week intervention
  The SART is a Go/No-Go task. In the SART, each digit is presented for 500 ms, followed by a mask presented for 900 ms (for a total trial duration of 5900 ms),260 trials in total. If no response was made to a go stimulus (the digits 1-2 and 4-9), this was coded as an omission. Responses to the no-go stimulus (3) were coded as errors. The question of randomly inserting 13 probes is to examine the current attention state of the subjects.
Weekly changes of The Subjective well-being scale during the intervention | pre-intervention; after the 3rd week intervention; after the 5rd week intervention; after the 7-week intervention
  The Subjective Well-being Scale is a self-reported questionnaire measuring individual's well-being level. Scores range from 0 to 35, with higher scores indicating higher levels of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — School of Psychological and Cognitive Sciences, Peking University
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No